CLINICAL TRIAL: NCT02364570
Title: Cardioprotective Activities Of Whole Eggs On Vascular Endothelial Function In Prediabetic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Richard Bruno, Associate Professor and Principal Investigator, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2014H0307; 2014H0307 (Other: Ohio State University IRB)
Record Dates: First submitted 2015-02-04; First posted 2015-02-18 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Prediabetes; Cardiovascular Disease
Keywords: CVD; Hyperglycemia; Postprandial; Vascular Function
MeSH Terms: conditions — Prediabetic State; Cardiovascular Diseases; Hyperglycemia | interventions — Glucose; Egg White; Egg Yolk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oral Glucose Tolerance Test (Active Comparator): We will perform fasting measurements of flow-mediated dilation (FMD) using ultrasound, and draw a blood sample, prior to administration of the test meal. Following these baseline measurements, participants will ingest glucose (100 g). FMD will be performed intermittently post-ingestion at 30, 60, 90, 120, 150, and 180 minutes. Blood samples will be collected at 0 min (immediately prior to eating) and at 30, 60, 90, 120, 150, and 180 minutes following the ingestion of the meal. After each blood sample is obtained, the catheter will be flushed with saline in order to prevent the formation of clots and to minimize the likelihood of having to insert a needle again. Subjects will remain supine in a comfortable position for the entire duration of the test.
  Interventions: Other: Glucose (100g)
- Glucose with Whole Eggs (Experimental): We will perform fasting measurements of flow-mediated dilation (FMD) using ultrasound, and draw a blood sample, prior to administration of the test meal. Following these baseline measurements, participants will ingest glucose (75 g) with 1.5 whole eggs (cooked). FMD will be performed intermittently post-ingestion at 30, 60, 90, 120, 150, and 180 minutes. Blood samples will be collected at 0 min (immediately prior to eating) and at 30, 60, 90, 120, 150, and 180 minutes following the ingestion of the meal. After each blood sample is obtained, the catheter will be flushed with saline in order to prevent the formation of clots and to minimize the likelihood of having to insert a needle again. Subjects will remain supine in a comfortable position for the entire duration of the test.
  Interventions: Other: Glucose (75g); Other: Whole Eggs
- Glucose with Egg Whites (Experimental): We will perform fasting measurements of flow-mediated dilation (FMD) using ultrasound, and draw a blood sample, prior to administration of the test meal. Following these baseline measurements, participants will ingest glucose (75 g) with 7 egg whites (cooked). FMD will be performed intermittently post-ingestion at 30, 60, 90, 120, 150, and 180 minutes. Blood samples will be collected at 0 min (immediately prior to eating) and at 30, 60, 90, 120, 150, and 180 minutes following the ingestion of the meal. After each blood sample is obtained, the catheter will be flushed with saline in order to prevent the formation of clots and to minimize the likelihood of having to insert a needle again. Subjects will remain supine in a comfortable position for the entire duration of the test.
  Interventions: Other: Glucose (75g); Other: Egg Whites
- Glucose with Egg Yolks (Experimental): We will perform fasting measurements of flow-mediated dilation (FMD) using ultrasound, and draw a blood sample, prior to administration of the test meal. Following these baseline measurements, participants will ingest glucose (75 g) with 2 egg yolks (cooked). FMD will be performed intermittently post-ingestion at 30, 60, 90, 120, 150, and 180 minutes. Blood samples will be collected at 0 min (immediately prior to eating) and at 30, 60, 90, 120, 150, and 180 minutes following the ingestion of the meal. After each blood sample is obtained, the catheter will be flushed with saline in order to prevent the formation of clots and to minimize the likelihood of having to insert a needle again. Subjects will remain supine in a comfortable position for the entire duration of the test.
  Interventions: Other: Glucose (75g); Other: Egg Yolks

INTERVENTIONS:
Other: Glucose (100g) — Ingestion of glucose (100g)
  Arms: Oral Glucose Tolerance Test
Other: Glucose (75g) — Ingestion of glucose (75g)
  Arms: Glucose with Egg Whites; Glucose with Egg Yolks; Glucose with Whole Eggs
Other: Whole Eggs — Ingestion of 1.5 whole eggs
  Arms: Glucose with Whole Eggs
Other: Egg Whites — Ingestion of 7 egg whites
  Arms: Glucose with Egg Whites
Other: Egg Yolks — Ingestion of 2 egg yolks
  Arms: Glucose with Egg Yolks

SUMMARY:
Cardiovascular disease (CVD) is largely a lifestyle-related condition that is the #1 killer of adults in the United States. Our work is aimed at understanding how short-term increases in blood sugar, like those that accompany eating a meal, affect blood vessel function and the risk of CVD. This research is aimed at understanding how meals composed of eggs affect short-term increases in blood sugar from eating, which are connected with increased risk of CVD. In particular, the investigators are trying to identify a specific meal composed of either whole eggs, egg yolks, or egg whites, that best reduces acute increases in blood sugar brought on by meals that consist of majority carbohydrate. At the same time, the investigators are trying to explore the protective affects that eggs may have on blood vessel function and the reduction of CVD risk.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in the United States [1]. The inability of your blood vessels to properly enlarge and shrink, known as vascular endothelial dysfunction (VED), is an early event leading to CVD and can be caused by postprandial hyperglycemia (PPH) [1] or short-term increases in blood sugar that occur after you have eaten. Although we do not know how this occurs, research shows that temporary increases in blood sugar impair the blood vessel's ability to properly enlarge and shrink. We also know that impaired vessel function is an early event leading to CVD and that research shows that short-term increases in blood sugar impair blood vessel function, even in healthy people [2].

Because high blood levels of cholesterol increase CVD risk, this has triggered flawed guidelines to restrict cholesterol in our diet [3], including limiting egg consumption. The misguided fear towards eating eggs has been routinely challenged by large-scale studies failing to associate eggs with heart disease risk [4-8]. Research shows that eggs improve the functioning of insulin to reduce blood sugar [9]. They also contain bioactive peptides that may attenuate oxidative stress [10-11]. This provides rationale for their study as a dietary strategy to reduce PPH and VED. Thus, the objective of this study is to define the potential benefits of eggs and its components (egg yolk and egg whites) on blood vessel health in adults with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

1. fasting glucose 100-125 mg/dL,
2. non-dietary supplement user,
3. no medications affecting vasodilation, inflammation, or energy metabolism,
4. no CVD,
5. nonsmokers,
6. individuals having blood pressure <130/85 mmHg and total cholesterol <240 mg/dL.

Exclusion Criteria:

1. unstable weight (±2 kg),
2. vegetarian or egg allergy,
3. alcohol intake >3 drinks/d or >10 drinks/wk), or
4. ≥7 h/wk of aerobic activity.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bruno, PhD, RD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):e28-e292. doi: 10.1161/01.cir.0000441139.02102.80. Epub 2013 Dec 18. No abstract available. PMID 24352519
- [Background] DECODE Study Group, the European Diabetes Epidemiology Group.. Glucose tolerance and cardiovascular mortality: comparison of fasting and 2-hour diagnostic criteria. Arch Intern Med. 2001 Feb 12;161(3):397-405. doi: 10.1001/archinte.161.3.397. PMID 11176766
- [Background] U.S. Dept of Agriculture and U.S. Dept of Health and Human Services (2010) Dietary Guidelines for Americans. 7th Ed.
- [Background] Djousse L, Gaziano JM. Egg consumption in relation to cardiovascular disease and mortality: the Physicians' Health Study. Am J Clin Nutr. 2008 Apr;87(4):964-9. doi: 10.1093/ajcn/87.4.964. PMID 18400720
- [Background] Hu Y, Liu W, Huang R, Zhang X. Postchallenge plasma glucose excursions, carotid intima-media thickness, and risk factors for atherosclerosis in Chinese population with type 2 diabetes. Atherosclerosis. 2010 May;210(1):302-6. doi: 10.1016/j.atherosclerosis.2009.11.015. Epub 2009 Nov 20. PMID 20005514
- [Background] Nakamura Y, Iso H, Kita Y, Ueshima H, Okada K, Konishi M, Inoue M, Tsugane S. Egg consumption, serum total cholesterol concentrations and coronary heart disease incidence: Japan Public Health Center-based prospective study. Br J Nutr. 2006 Nov;96(5):921-8. doi: 10.1017/bjn20061937. PMID 17092383
- [Background] Sauvaget C, Nagano J, Allen N, Grant EJ, Beral V. Intake of animal products and stroke mortality in the Hiroshima/Nagasaki Life Span Study. Int J Epidemiol. 2003 Aug;32(4):536-43. doi: 10.1093/ije/dyg151. PMID 12913025
- [Background] Scrafford CG, Tran NL, Barraj LM, Mink PJ. Egg consumption and CHD and stroke mortality: a prospective study of US adults. Public Health Nutr. 2011 Feb;14(2):261-70. doi: 10.1017/S1368980010001874. Epub 2010 Jul 16. PMID 20633314
- [Background] Blesso CN, Andersen CJ, Barona J, Volek JS, Fernandez ML. Whole egg consumption improves lipoprotein profiles and insulin sensitivity to a greater extent than yolk-free egg substitute in individuals with metabolic syndrome. Metabolism. 2013 Mar;62(3):400-10. doi: 10.1016/j.metabol.2012.08.014. Epub 2012 Sep 27. PMID 23021013
- [Background] Davalos A, Miguel M, Bartolome B, Lopez-Fandino R. Antioxidant activity of peptides derived from egg white proteins by enzymatic hydrolysis. J Food Prot. 2004 Sep;67(9):1939-44. doi: 10.4315/0362-028x-67.9.1939. PMID 15453585
- [Background] Nimalaratne C, Lopes-Lutz D, Schieber A, Wu J. Effect of domestic cooking methods on egg yolk xanthophylls. J Agric Food Chem. 2012 Dec 26;60(51):12547-52. doi: 10.1021/jf303828n. Epub 2012 Dec 14. PMID 23205520
- [Background] McDonald JD, Chitchumroonchokchai C, Li J, Mah E, Labyk AN, Reverri EJ, Ballard KD, Volek JS, Bruno RS. Replacing carbohydrate during a glucose challenge with the egg white portion or whole eggs protects against postprandial impairments in vascular endothelial function in prediabetic men by limiting increases in glycaemia and lipid peroxidation. Br J Nutr. 2018 Feb;119(3):259-270. doi: 10.1017/S0007114517003610. Epub 2018 Jan 16. PMID 29335039
- [Background] McDonald JD, Mah E, Chitchumroonchokchai C, Reverri EJ, Li J, Volek JS, Villamena FA, Bruno RS. Co-ingestion of whole eggs or egg whites with glucose protects against postprandial hyperglycaemia-induced oxidative stress and dysregulated arginine metabolism in association with improved vascular endothelial function in prediabetic men. Br J Nutr. 2018 Oct;120(8):901-913. doi: 10.1017/S0007114518002192. Epub 2018 Aug 30. PMID 30160222

RESULTS

PARTICIPANT FLOW:
Groups:
- Glucose, Then Whole Egg, Then Egg White, Then Egg Yolk; Glucose, Then Egg White, Then Whole Egg, Then Egg Yolk; Glucose, Then Egg Yolk, Then Egg White, Then Whole Egg; Glucose, Then Whole Egg, Then Egg Yolk, Then Egg White; Glucose, Then Egg White, Then Egg Yolk, Then Whole Egg; Whole Egg, Then Egg White, Then Egg Yolk, Then Glucose; Whole Egg, Then Egg Yolk, Then Egg White, Then Glucose; Whole Egg, Then Glucose, Then Egg Yolk, Then Egg White; Egg White, Then Glucose, Then Whole Egg, Then Egg Yolk; Egg White, Then Egg Yolk, Then Whole Egg, Then Glucose; Whole Egg, Then Glucose, Then Egg White, Then Egg Yolk; Egg Yolk, Then Egg White, Then Whole Egg, Then Glucose; Egg Yolk, Then Whole Egg, Then Glucose, Then Egg White; Egg Yolk, Then Glucose, Then Egg White, Then Whole Egg; Egg Yolk, Then Egg White, Then Glucose, Then Whole Egg: We will perform fasting measurements of flow-mediated dilation (FMD) using ultrasound, and draw a blood sample, prior to administration of the test meal. Following these baseline measurements, participants will ingest glucose (100 g), or glucose (75 g) + 1.5 cooked whole eggs, or glucose (75 g) + 7 egg whites, or glucose (75 g) + 2 egg yolks. FMD will be performed intermittently post-ingestion at 30, 60, 90, 120, 150, and 180 minutes. Blood samples will be collected at 0 min (immediately prior to eating) and at 30, 60, 90, 120, 150, and 180 minutes following the ingestion of the meal.
- Glucose, Then Egg Yolk, Then Whole Egg, Then Egg White: We will perform fasting measurements of flow-mediated We will perform fasting measurements of flow-mediated dilation (FMD) using ultrasound, and draw a blood sample, prior to administration of the test meal. Following these baseline measurements, participants will ingest glucose (100 g), or glucose (75 g) + 1.5 cooked whole eggs, or glucose (75 g) + 7 egg whites, or glucose (75 g) + 2 egg yolks. FMD will be performed intermittently post-ingestion at 30, 60, 90, 120, 150, and 180 minutes. Blood samples will be collected at 0 min (immediately prior to eating) and at 30, 60, 90, 120, 150, and 180 minutes following the ingestion of the meal.
Period: Overall Study
Arm/Group | Glucose, Then Whole Egg, Then Egg White, Then Egg Yolk | Glucose, Then Egg White, Then Whole Egg, Then Egg Yolk | Glucose, Then Egg Yolk, Then Egg White, Then Whole Egg | Glucose, Then Egg Yolk, Then Whole Egg, Then Egg White | Glucose, Then Whole Egg, Then Egg Yolk, Then Egg White | Glucose, Then Egg White, Then Egg Yolk, Then Whole Egg | Whole Egg, Then Egg White, Then Egg Yolk, Then Glucose | Whole Egg, Then Egg Yolk, Then Egg White, Then Glucose | Whole Egg, Then Glucose, Then Egg Yolk, Then Egg White | Egg White, Then Glucose, Then Whole Egg, Then Egg Yolk | Egg White, Then Egg Yolk, Then Whole Egg, Then Glucose | Whole Egg, Then Glucose, Then Egg White, Then Egg Yolk | Egg Yolk, Then Egg White, Then Whole Egg, Then Glucose | Egg Yolk, Then Whole Egg, Then Glucose, Then Egg White | Egg Yolk, Then Glucose, Then Egg White, Then Whole Egg | Egg Yolk, Then Egg White, Then Glucose, Then Whole Egg
Started | 1 | 1 | 2 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 1 | 1 | 2 | 1 | 1
Completed | 1 | 1 | 2 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 1 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants received all 4 interventions in a randomized order (Oral Glucose Tolerance Test, Glucose with Whole Eggs, Glucose with Egg Whites, Glucose with Egg Yolks). We will perform fasting measurements of flow-mediated dilation (FMD) using ultrasound, and draw a blood sample, prior to administration of the test meal. FMD will be performed intermittently post-ingestion of the test meal at 30, 60, 90, 120, 150, and 180 minutes. Blood samples will be collected at 0 min (immediately prior to eating) and at 30, 60, 90, 120, 150, and 180 minutes following the ingestion of the meal. After each blood sample is obtained, the catheter will be flushed with saline in order to prevent the formation of clots and to minimize the likelihood of having to insert a needle again. Subjects will remain supine in a comfortable position for the entire duration of the test.
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.1 (2.5)
Fasting Glucose [Mean (Standard Deviation); unit: mmol/L] | 6.0 (0.4)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.0 (0.6)
Insulin [Mean (Standard Deviation); unit: pmol/L] | 144.8 (15.8)
Triglyceride [Mean (Standard Deviation); unit: mmol/L] | 1.5 (0.6)
HDL Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 0.64 (0.16)
LDL Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 3.7 (0.8)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 123 (6)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 72 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Vascular Endothelial Function
Description: Flow mediated dilation (FMD) evaluated on the basis as change from baseline to calculate FMD area under the curve from 0-180 min, i.e. i.e. Area Under the Curve (AUC) of change from baseline in FMD from 0 min to 180 min (i.e., AUC (FMD 0 min- 0 min, FMD 30 min-0 min, FMD 60 min-0 min, etc)
Time Frame: Area under the curve of brachial artery FMD for 3 hours (0, 30, 60, 90, 120 min)
Measure: Mean (Standard Error); unit: %FMD*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
%FMD*min | -294.4 (41.35) | -152.9 (36.9) | -102.9 (34.31) | -361.6 (48.55)

2. Secondary Outcome: Glucose
Description: Glucose concentrations evaluated on the basis as change from baseline to calculate glucose area under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in glucose from 0 min to 180 min (i.e., AUC (glucose 0 min- 0 min, glucose 30 min-0 min, glucose 60 min-0 min, etc)
Time Frame: Area under the curve for plasma glucose for 3 hours (0, 30, 60, 90, 120 min)
Measure: Mean (Standard Error); unit: mmol/L*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
mmol/L*min | 461.9 (77.78) | 247.5 (52.67) | 296.1 (61.16) | 390.6 (51.13)

3. Secondary Outcome: Oxidative Stress Biomarker (Malondialdehyde; MDA)
Description: MDA concentrations evaluated on the basis as change from baseline to calculate MDAarea under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in MDA from 0 min to 180 min (i.e., AUC (MDA 0 min- 0 min, MDA 30 min-0 min, MDA 60 min-0 min, etc)
Time Frame: Area under curve of MDA for 3 hours (0, 30, 60, 90, 120, 150, 180 min)
Measure: Mean (Standard Error); unit: umol/L*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
umol/L*min | 52.97 (8.674) | 16.51 (8.978) | 30.04 (4.996) | 59.2 (3.728)

4. Secondary Outcome: Insulin
Description: Insulin concentrations evaluated on the basis as change from baseline to calculate insulin area under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in insulin from 0 min to 180 min (i.e., AUC (Insulin 0 min- 0 min, insulin 30 min-0 min, insulin 60 min-0 min, etc)
Time Frame: Area under the curve for plasma insulin for 3 hours (0, 30, 60, 90, 120 min)
Measure: Mean (Standard Error); unit: mmol/L*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
mmol/L*min | 99433 (14623) | 73970 (14917) | 72645 (15709) | 79235 (16634)

5. Secondary Outcome: Cholecystokinin (CCK)
Description: CCK concentrations evaluated on the basis as change from baseline to calculate CCK area under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in CCK from 0 min to 180 min (i.e., AUC (CCK 0 min- 0 min, CCK 30 min-0 min, CCK 60 min-0 min, etc)
Time Frame: Area under the curve for 3 hours (0, 30, 60, 90, 120 minutes)
Measure: Mean (Standard Error); unit: pmol/L*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
pmol/L*min | -254.018 (54.122) | 93.659 (72.540) | -29.193 (80.656) | -150.550 (78.186)

6. Secondary Outcome: Methylglyoxal (MGO)
Description: MGO concentrations evaluated on the basis as change from baseline to calculate MGO area under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in MGO from 0 min to 180 min (i.e., AUC (MGO 0 min- 0 min, MGO 30 min-0 min, MGO 60 min-0 min, etc)
Time Frame: Area under the curve for methylglyoxal for 3 hours (0, 30, 60, 90, 120 min)
Measure: Mean (Standard Error); unit: nmol/L*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
nmol/L*min | 2318.9 (394.61) | 1807.4 (264.49) | 1742.3 (244.57) | 2611.8 (229.58)

7. Secondary Outcome: 8-isoprostaglandin-F2a
Description: 8-isoprostaglandin-F2a concentrations evaluated on the basis as change from baseline to calculate 8-isoprostaglandin-F2a area under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in 8-isoprostaglandin-F2a from 0 min to 180 min (i.e., AUC (8-isoprostaglandin-F2a 0 min- 0 min, 8-isoprostaglandin-F2a 30 min-0 min, 8-isoprostaglandin-F2a 60 min-0 min, etc)
Time Frame: Area under the curve for 8-isoprostaglandin-F2a for 3 hours (0, 30, 60, 90, 120 min)
Measure: Mean (Standard Error); unit: pmol/L*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
pmol/L*min | 767110 (187143) | 306758 (185617) | 39117 (90562) | 718932 (199003)

8. Secondary Outcome: Arachidonic Acid (AA)
Description: Arachidonic acid concentrations evaluated on the basis as change from baseline to calculate arachidonic acid area under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in arachidonic acid from 0 min to 180 min (i.e., AUC (arachidonic acid 0 min- 0 min, arachidonic acid 30 min-0 min, arachidonic acid 60 min-0 min, etc)
Time Frame: Area under the curve for arachidonic acid for 3 hours (0, 30, 60, 90, 120 min)
Measure: Mean (Standard Error); unit: umol/L*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
umol/L*min | -4771.6 (2971.8) | -6408.8 (2519.3) | -6109.1 (3093.4) | -10354 (3273.3)

9. Secondary Outcome: 8-isoprostaglandin-F2a/Arachidonic Acid
Description: 8-isoprostaglandin-F2a/arachidonic acid concentrations evaluated on the basis as change from baseline to calculate 8-isoprostaglandin-F2a/arachidonic acid area under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in 8-isoprostaglandin-F2a/arachidonic acid from 0 min to 180 min (i.e., AUC (8-isoprostaglandin-F2a/arachidonic acid 0 min- 0 min, 8-isoprostaglandin-F2a/arachidonic acid 30 min-0 min, 8-isoprostaglandin-F2a/arachidonic acid 60 min-0 min, etc)
Time Frame: Area under the curve for 8-isoprostaglandin-F2a/arachidonic acid for 3 hours (0, 30, 60, 90, 120 min)
Measure: Mean (Standard Error); unit: (pmol/L)/(umol/L)*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
(pmol/L)/(umol/L)*min | 1254.6 (263.54) | 435.70 (141.32) | 538.81 (100.61) | 1151.2 (255.58)

10. Secondary Outcome: Nitric Oxide Metabolites (Nitrites/Nitrates) (NOx)
Description: Biomarker of nitric oxide homeostasis is based on the assessment of total nitrite and nitrate concentrations. Changes relative to baseline were used to calculate area under the curve of total nitric oxide metabolites from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in nitric oxide homeostasis from 0 min to 180 min (i.e., AUC (NOx 0 min- 0 min, NOx 30 min-0 min, NOx 60 min-0 min, etc)
Time Frame: Area under the curve for NOx for 3 hours (0, 30, 60, 90, 120 min)
Measure: Mean (Standard Error); unit: umol/L*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
umol/L*min | -1213.9 (231.31) | -39.71 (277.07) | -245.34 (225.96) | 607.12 (315.01)

11. Secondary Outcome: Arginine (Arg)
Description: Arginine concentrations evaluated on the basis as change from baseline to calculate arginine area under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in arginine from 0 min to 180 min (i.e., AUC (arginine 0 min- 0 min, arginine 30 min-0 min, arginine 60 min-0 min, etc)
Time Frame: Area under the curve for arginine for 3 hours (0, 30, 60, 90, 120 min)
Measure: Mean (Standard Error); unit: umol/L*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
umol/L*min | -3645.2 (313.94) | -1714.4 (227.65) | 503.67 (506.09) | -1472.5 (407.00)

12. Secondary Outcome: Asymmetric Dimethylarginine/Arginine (ADMA/Arg)
Description: ADMA/Arg concentrations evaluated on the basis as change from baseline to calculate ADMA/Arg area under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in ADMA/Arg from 0 min to 180 min (i.e., AUC (ADMA/Arg 0 min- 0 min, ADMA/Arg 30 min-0 min, ADMA/Arg 60 min-0 min, etc)
Time Frame: Area under the curve for ADMA/Arg for 3 hours (0, 30, 60, 90, 120 min)
Measure: Mean (Standard Error); unit: (nmol/L)/(umol/L)*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
(nmol/L)/(umol/L)*min | 195.86 (29.75) | 59.30 (22.83) | -44.04 (21.57) | 118.62 (23.36)

13. Secondary Outcome: Symmetric Dimethylarginine/Arginine (SDMA/Arg)
Description: SDMA/Arg concentrations evaluated on the basis as change from baseline to calculate SDMA/Arg area under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in SDMA/Arg from 0 min to 180 min (i.e., AUC (SDMA/Arg 0 min- 0 min, SDMA/Arg 30 min-0 min, SDMA/Arg 60 min-0 min, etc)
Time Frame: Area under the curve for SDMA/Arg for 3 hours (0, 30, 60, 90, 120 min)
Measure: Mean (Standard Error); unit: (nmol/L)/(umol/L)*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
(nmol/L)/(umol/L)*min | 178.48 (17.19) | 62.43 (17.50) | -37.95 (18.72) | 86.03 (11.88)

14. Secondary Outcome: Angiotensin-II
Description: Angiotensin-II concentrations evaluated on the basis as change from baseline to calculate angiotensin-II area under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in angiotensin-II from 0 min to 180 min (i.e., AUC (angiotensin-II 0 min- 0 min, angiotensin-II 30 min-0 min, angiotensin-II 60 min-0 min, etc)
Time Frame: Area under the curve for angiotensin-II for 3 hours (0, 30, 60, 90, 120 min)
Measure: Mean (Standard Error); unit: pg/mL*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
pg/mL*min | 1223.0 (146.47) | 292.45 (55.01) | 316.19 (51.09) | 341.89 (59.04)

15. Secondary Outcome: Endothelin-I
Description: Endothelin-I concentrations evaluated on the basis as change from baseline to calculate endothelin-I area under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in endothelin-I from 0 min to 180 min (i.e., AUC (endothelin-I 0 min- 0 min, endothelin-I 30 min-0 min, endothelin-I 60 min-0 min, etc)
Time Frame: Area under the curve for endothelin-I for 3 hours (0, 30, 60, 90, 120 min)
Measure: Mean (Standard Error); unit: pg/mL*min
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Number analyzed (Participants) | 20 | 20 | 20 | 20
pg/mL*min | 27.08 (7.03) | -13.29 (10.32) | -1.97 (11.29) | 5.59 (10.08)

ADVERSE EVENTS:
Time Frame: Participants were monitored for any adverse events in response to a glucose challenge in the absence or presence of egg-based meals through study completion (~6 total weeks).
Arm/Group | Oral Glucose Tolerance Test | Glucose With Whole Eggs | Glucose With Egg Whites | Glucose With Egg Yolks
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
This study replaced carbohydrate in a glucose challenge with isocaloric amounts of whole eggs, egg whites, and egg yolks. Future studies should consider equi-carbohydrate based meals with or without equal portions of egg components.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No